CLINICAL TRIAL: NCT03120702
Title: Measurement of Total Hemoglobin by Pulse Oximetry in Neonatal Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: CHOC0002
Record Dates: First submitted 2017-04-14; First posted 2017-04-19 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Neonatal Test Subjects (Experimental): All test subjects in this group are neonatal patients who will receive a investigational Rainbow SpHb sensor.
  Interventions: Device: Investigational Rainbow SpHb sensor

INTERVENTIONS:
Device: Investigational Rainbow SpHb sensor — Investigational Rainbow SpHb sensor

SUMMARY:
Assess ability of Masimo SpHb sensor to demonstrate robust performance on various sensor application sites on neonates/infants

ELIGIBILITY:
Inclusion Criteria:

* Male or female newborn infants of any gestational age requiring at least one (1) blood draw as part of their routine care.
* Ages: Newborn infants less than 16 weeks postnatal age.
* Weight: Range from 500 g to 10 kg.
* Able to obtain written informed consent from parents or legal guardians

Exclusion Criteria:

* Neonatal patients with abnormalities at the planned application sites that would interfere with transilluminating the foot or hand like unusual deformities of limbs, absence of feet, severe edema, localized infections, and other.

Max Age: 16 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2013-07-23 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

PRIMARY OUTCOMES:
Assess ability of Masimo SpHb sensor to demonstrate robust performance on various sensor application sites on neonates/infants | duration of surgery
  To study the SpHb sensor in neonatal population.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Orange County, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No